CLINICAL TRIAL: NCT00529633
Title: Phase 3 Study: The Effect of Thalidomide in Suppression of the Systemic Inflammatory Response Syndrome in Hemodialysis Patients
Brief Title: The Effect of Thalidomide in Suppression of the Systemic Inflammatory Response Syndrome in Hemodialysis Patients
Acronym: ICM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment -- We could not recruit patients willing to be enrolled
Sponsor: George A. Kaysen, M.D. (Other)
Collaborators: Beth Israel Medical Center (Other)
Responsible Party: Sponsor-Investigator, George A. Kaysen, M.D., Professor of Medicine, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200614929
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Hypoalbuminemia
Keywords: Inflammation; albumin
MeSH Terms: conditions — Hypoalbuminemia; Inflammation | interventions — Thalidomide; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide (Active Comparator): 1. 12 End stage renal disease (ESRD) patients on hemodialysis for at least 3 months
  2. Serum C reactive protein level of ≥ 0.8 mg/dl
  3. Serum albumin < 3.8 g/dl (BCG)
  4. Patients will receive 100mg Thalidomide for a period of 4 weeks; if somnolence tolerated, dosage is increased to 200mg nightly for a period of 20 more weeks -- to total of 24 weeks on Thalidomide.
  Interventions: Drug: Thalidomide
- No Drug (Placebo Comparator): 1. 12 End stage renal disease (ESRD) patients on hemodialysis for at least 3 months
  2. Serum C reactive protein level of ≥ 0.8 mg/dl
  3. Serum albumin < 3.8 g/dl (BCG)
  4. Patients will receive Placebo (Sugar pill) for a period of 24 weeks.
  Interventions: Other: Sugar pill

INTERVENTIONS:
Drug: Thalidomide — Thalidomide by mouth at night for a total of 24 weeks
  Arms: Thalidomide
Other: Sugar pill — Placebo by mouth at night for a total of 24 weeks
  Other Names: Placebo (no drug)
  Arms: No Drug

SUMMARY:
Both malnutrition and inflammation are associated with death in dialysis patients and also with cardiovascular disease. The researchers are testing the idea that inflammation causes malnutrition by using a drug to suppress inflammation in hemodialysis patients to find out whether that will increase blood tests that are associated with malnutrition. The researchers will give hemodialysis patients who have both inflammation and malnutrition either thalidomide or a placebo and compare the effects of treatment on the levels of two proteins in the blood, albumin and prealbumin, that are normally reduced in malnourished patients. Patients who have a serum albumin concentration < 3.8 g/dl will be asked to sign consent to have blood drawn prior to dialysis for measurement of CRP (C-reactive protein). Those with CRP values ≥ 0.8 mg/dl will have a second measurement of CRP performed within 2 weeks. Those with two consecutive values of CRP ≥ 0.8 mg/dl will be eligible for enrollment

DETAILED DESCRIPTION:
4.1 Pre-assignment measurements will include:

1. Patient is eligible for enrollment.
2. Complete physical examination.
3. Blood draw at initiation of hemodialysis session
4. Instruction on birth control methods required.
5. Subjects who are non-compliant with regard to medication compliance range or birth control requirements as outlined in the S.T.E.P.S.® program will be immediately discontinued from the study

4.2 Detailed description of treatment: Patients who completed the first 4 weeks will be randomized into Treatment group. A total of 24 subjects will be studied; 12 will receive no drug and 12 will receive thalidomide. Subjects randomized to "Active" Treatment arm will receive Placebo (no-drug/sugar pill) ,or thalidomide 100 mg (two 50 mg active capsules) to take at bedtime. Weekly, Subjects will have blood drawn; will undergo a capsule count to establish a compliance range of > 85%; will have physical exam with special attention to skin and evaluation of peripheral nervous system for a change in or appearance of sensory neuropathy.

If somnolence is tolerable (subjects do not have residual somnolence in the morning) the dose will be increased to 200 mg (4 capsules).

Patients who completed 24 weeks of study will have final evaluation at week 28.

ELIGIBILITY:
Inclusion Criteria:

1. End stage renal disease (ESRD) patients on hemodialysis for at least 3 months.
2. Serum C reactive protein level of ≥ 0.8 mg/dl.
3. Serum albumin < 3.8 g/dl (BCG).
4. Signing a written informed consent form.
5. Willingness and ability to comply with the FDA-mandated S.T.E.P.S ® program.
6. Age > 18 years.

Exclusion Criteria:

1. Pregnant and/ or lactating female.
2. Active infection within the previous 8 weeks requiring administration of antibiotics.
3. Patients receiving systemic immunosuppressive therapy.
4. Patients with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Kaysen, MD Ph.D, Principal Investigator — University of California, Davis; James F. Winchester, MD, Study Director — Beth Israel Medicial Center New York New York
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been terminated due to lack of participation. We enrolled 16 subjects according to eligibility. 4 subjects randomized into the study. Two subjects completed the study.
Pre-assignment Details: Subject enrollment into the "active" study must meet capsule count of >85% compliance with regard to medication and/or birth control requirements as outlined in the S.T.E.P.S ® in the first 4 weeks of study program
Groups:
- Placebo: This arm will consist of hemodialysis patients having elevated CRP and low albumin levels (less than 3.8 by BCG) who will be treated with a placebo for 24 weeks.
  Blood will be drawn every 4 weeks for measurement of CRP, albumin and prealbumin. Subject must meet capsule count of >85% compliance with regard to medication and/or birth control requirements as outlined in the S.T.E.P.S ® in the first 4 weeks of study program
- Thalidomide: 1. End stage renal disease (ESRD) patients on hemodialysis for at least 3 months
  2. Serum C reactive protein level of ≥ 0.8 mg/dl
  3. Serum albumin < 3.8 g/dl (BCG)
  4. Patients will receive Thalidomide for a period of 24 weeks.
  5. Blood will be drawn every 4 weeks for a total of 28 weeks to establish the effect on albumin, prealbumin and CRP
  Thalidomide : 100 mg by mouth at night for 4 weeks 200 mg by mouth at night for 20 weeks
Period: Overall Study
Arm/Group | Placebo | Thalidomide
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Thalidomide: 1. 12 End stage renal disease (ESRD) patients on hemodialysis for at least 3 months
  2. Serum C reactive protein level of ≥ 0.8 mg/dl
  3. Serum albumin < 3.8 g/dl (BCG)
  4. Patients will receive Thalidomide for a period of 24 weeks.100 mg by mouth at night for 4 weeks; then if tolerated, Thalidomid will be increased to 200 mg by mouth at night for 20 weeks; for a total of 24 weeks on Thalidomid
- Placebo: 1. 12 End stage renal disease (ESRD) patients on hemodialysis for at least 3 months
  2. Serum C reactive protein level of ≥ 0.8 mg/dl
  3. Serum albumin < 3.8 g/dl (BCG)
  4. Patients will receive Placebo for a period of 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Thalidomide | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Difference in Serum Albumin
Description: Serum albumin in treated patient and control ("no drug") patients were tabulated once weekly for week #1-4 , then once every 4 weeks thereafter at week# 8, 12, 16, 20, 24 to see changes of health status. Final data collected at week 28 -- to ensure patient safety
Time Frame: 28 weeks total
Measure: Number; unit: g/dL of Albumin
Groups:
- Thalidomide: This arm will consist of hemodialysis patients having elevated CRP and low albumin levels (less than 3.8 by BCG) who will be treated with Thalidomide for 24 weeks. Blood will be drawn every 4 weeks for measurement of CRP, albumin and prealbumin Dosage at 2x 50mg each night; if somnolence tolerated, dosage will increase to 4x50mg per night
- Placebo: Placebo Control--This arm will consist of hemodialysis patients having elevated CRP and low albumin levels (less than 3.8 by BCG) who will be treated with a placebo for 24 weeks. Blood will be drawn every 4 weeks for measurement of CRP, albumin and prealbumin
Arm/Group | Thalidomide | Placebo
Number analyzed (Participants) | 1 | 1
g/dL of Albumin
  week 1 | 3.4 | 3.7
  week 2 | 3.7 | 3.5
  week 3 | 3.5 | 3.4
  week 4 | 3.6 | 4.0
  week 8 | 3.8 | 3.6
  week 12 | 3.6 | 4.1
  week 16 | 3.5 | 4.0
  week 20 | 2.9 | 3.8
  week 24 | 3.6 | 3.9
  week 28 | 3.5 | 3.9

2. Primary Outcome: Difference in Serum CRP
Description: Serum CRP in treated patient and control ("no drug") patients were tabulated once weekly for week #1-4 , then once every 4 weeks thereafter at week# 8, 12, 16, 20, 24 to see changes of health status. Final data collected at week 28 -- to ensure patient safety
Time Frame: 28 weeks total
Measure: Number; unit: Mg/L CRP
Arm/Group | Thalidomide | Placebo
Number analyzed (Participants) | 1 | 1
Mg/L CRP
  week 1 | NA — Observation below quantifiable range | 1.76
  week 2 | NA — Observation above quantifiable range | 2.07
  week 3 | NA — Observation below quantifiable range | 1.76
  week 4 | NA — Observation below quantifiable range | 2.29
  week 8 | NA — Observation below quantifiable range | 2.87
  week 12 | NA — Observation above quantifiable range | 2.87
  week 16 | NA — Observation below quantifiable range | 3.41
  week 20 | NA — Observation above quantifiable range | 1.92
  week 24 | NA — Observation above quantifiable range | 6.01
  week 28 | NA — Observation below quantifiable range | 3.93

3. Primary Outcome: Difference in Serum Prealbumin
Description: Serum Prealbumin in treated patient and control ("no drug") patients were tabulated once weekly for week #1-4 , then once every 4 weeks thereafter at week# 8, 12, 16, 20, 24 to see changes of health status. Final data collected at week 28 -- to ensure patient safety
Time Frame: 28 weeks total
Population: Participant data is not available due to no shipping of specimen to analyzing laboratory
Arm/Group | Thalidomide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: weekly up to 24 weeks of active study period
Description: Adverse Event questionnaire was assessed at weekly visit
Groups:
- Thalidomide: Patients will receive Thalidomide for a period of 24 weeks. Blood will be drawn every 4 weeks for a total of 28 weeks to establish the effect on albumin, prealbumin and CRP.
  Thalidomide : 100 mg by mouth at night for 4 weeks; 200 mg by mouth at night for 20 weeks
- Placebo: This arm will consist of hemodialysis patients having elevated CRP and low albumin levels (less than 3.8 by BCG) who will be treated with a placebo for 24 weeks.
Arm/Group | Thalidomide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination -- Study is terminated due to low enrollment of subjects willing to enter this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No